CLINICAL TRIAL: NCT00294541
Title: An Open-Label Extension Study Evaluating the Long-Term Safety of ICA-17043 With or Without Hydroxyurea Therapy in Subjects With Sickle Cell Disease
Brief Title: A Study Evaluating the Long-Term Safety of ICA-17043 in Sickle Cell Disease Patients With or Without Hydroxyurea Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy demonstrated in study ICA-17043-10
Sponsor: Icagen (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICA-17043-12
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2007-09-11 (Estimated); Status verified 2007-09

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia
Keywords: sickle cell disease; sickle cell anemia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — senicapoc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: ICA-17043

SUMMARY:
This trial is a follow-up companion study to Protocol ICA-17043-10, a Phase III, multi-center, efficacy and safety study of ICA-17043. This is an open-label extension study collecting safety data on the use of ICA-17043 in subjects with sickle cell disease (SCD) (e.g., HbSS, HbSC, HbSb0-thalassemia, HbSb+-thalassemia subjects). All subjects who have successfully completed ICA-17043-10 will, if deemed appropriate by their study Investigator and appropriate consent by subject is given, enroll in the ICA-17043-12 study (Study 12). Only patients who participated in ICA-17043-10 are eligible for this open label study

ELIGIBILITY:
Inclusion Criteria:

* Successfully completed Study ICA-17043-10
* Discontinued Study 10 or 12 following the DMC recommendations because he/she was not on HU, and has since been on a stable dose of HU for at least 3 months prior to Day 1
* Male, or female not capable of becoming pregnant or using appropriate birth control
* Has willingly given written informed consent to participate in this study

Exclusion Criteria:

* The subject, if female, has a positive urine pregnancy test on Day 1 (before entering study)
* The subject is presently unsuitable for participation in this long-term study

Ages: 17 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-02; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Safety measures only | at least 60 weeks
No efficacy outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Stocker, PhD, Study Director — Icagen
Locations (31):
- United States (31):
  - University of South Alabama, Mobile, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Oakland, Oakland, California
  - University of California Davis Medical Center, Sacramento, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Century Clinical Research, Inc., Holly Hill, Florida
  - University of Florida Health Science Center, Jacksonville, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Illinois Medical Center, Chicago, Illinois
  - Sickle Cell Center of Northern Louisiana, Shreveport, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Wayne State School of Medicine, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Robert Wood Johnson Medical Center, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Medical College of Virginia, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia